CLINICAL TRIAL: NCT01053884
Title: Anidulafungin in Patients With Hematologic Malignancies - An Open-label, Prospective Study to Evaluate the Safety Profile at Prophylactic and Therapeutic Dosages
Brief Title: Anidulafungin in Patients With Hematologic Malignancies
Acronym: ECALTA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: reduced recruitment rate due to non infectious, but competitive trials at our institution
Sponsor: Elisabethinen Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Michael Girschikofsky, OA Dr. Michael Girschikofsky, Elisabethinen Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Anidulafungin - MG-ECALTA1; 2009-014527-23 (Other: EudraCT)
Record Dates: First submitted 2010-01-15; First posted 2010-01-22 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2009-07

CONDITIONS: Hematologic Malignancies
Keywords: Invasive Candidiasis; invasive fungal disease; Anidulafungin
MeSH Terms: conditions — Hematologic Neoplasms; Candidiasis, Invasive; Invasive Fungal Infections | interventions — Anidulafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anidulafungin, safety, antifungal drug (Other): single arm study
  Interventions: Drug: Anidulafungin

INTERVENTIONS:
Drug: Anidulafungin — standard dose: 200mg/d on day 1, followed by 100mg/d from day 2 as maintenance dose.
  Prophylaxis will be given until the recovery from neutropenia (ANC > 1,0 G/L without myelosupportive medications) and in cases of active fungal infection until best response, in case of fungemia for at least 2 weeks after the first negative culture.
  Other Names: Ecalta

SUMMARY:
Study objectives To evaluate the safety of the echinocandin anidulafungin for prophylaxis or treatment of invasive fungal infections (IFI) in hematologic patients.

Study design, Study conduct period Prospective, open label, phase II, one arm, single centre study October 2009 - September 2010

Study population Twenty adult patients (≥ 18 years) with a hematologic disorder and an indication for antifungal prophylaxis or therapy, but a relative contraindication for azoles or polyenes due to hepatic and renal dysfunction respectively

Methods and Main Out-come Variables Main Outcome Parameter Safety: Adverse events and changes of important laboratory parameters with clinical impact will be reported.

Secondary Outcome Parameter Efficacy: In therapeutically use the outcome will be categorized into success or failure. For patients receiving anidulafungin as prophylaxis the number and rate of breakthrough infections will be documented.

Risk assessment Treatment related adverse effects as reported in the approved physician prescribing information (usually mild and with an incidence of < 5%). Treatment failure due to resistant pathogens.

Expected benefit from this study IFI is a major cause of death among hematological patients, especially those undergoing high dose chemotherapy. It is conceivable that anidulafungin is a new treatment option for patients in whom azoles or polyenes are relatively contraindicated.

DETAILED DESCRIPTION:
Treatment of patients with hematologic disorders is frequently complicated by invasive fungal infections (IFI). The current spectrum of pathogens in this patient population is characterised by an increasing rate of aspergillosis, atypical moulds and yeasts, which might be explained by an extended application of myelosuppressive chemotherapy and prophylactic use of antibiotic therapy, but also more sensitive diagnostic tools. Although several new antifungal drugs have been approved recently for the treatment of invasive fungal infections, the mortality rates remain unacceptably high. In patients with suspected IFI invasive diagnostic procedures can often not be performed due to thrombocytopenia and blood testing of fungal antigens with ELISA or PCR-methods are at most additive tools at this time. Thus, antifungal drugs are frequently applied empirically when neutropenic fever persists despite of antibiotic therapy or preemptive in case of radiological or laboratory suspicion of IFI. The antifungal armamentarium consists mainly of azoles, polyenes, and echinocandins. Therapy with azoles is frequently complicated by hepatological side effects and drug interactions, whereas the application of polyenes is often associated with a worsening of the renal function, severe hypopotassemia and shivering. Because of their favourable efficacy and outstanding safety profile, nowadays echinocandins are increasingly used in hematologic wards, especially in patients with renal or liver comorbidity. Anidulafungin is a novel echinocandin with potent invitro fungicidal activity against several pathogen yeasts and moulds like Candida- or Aspergillus spp. It has recently been approved by the EMEA for treatment of invasive candidiasis in non-neutropenic patients. A low cytochrome P450 interaction profile has been reported and dose adaption in case of hepatical or renal impairment is not recommended. In the pivotal clinical trial anidulafungin achieved a superior response rate for treatment of invasive candida infection in comparison with fluconazole. In this trial, only a quarter of patients had cancer and only 3% had neutrophil counts below 500/cm3 blood at randomisation. Although the clinical experience of the efficacy and tolerability of anidulafungin in adult hematologic patients is limited, the Infectious Diseases Society of America recently recommended anidulafungin for use in neutropenic patients with candidiasis.

Primary endpoint:

Safety: For all patients who will receive anidulafungin without regard to indication the incidence of (serious) adverse events and changes of important laboratory parameters (in particular liver and renal function parameters) with clinical impact will be reported.

Secondary endpoints:

Pharmacokinetics Efficacy

For patients receiving anidulafungin as prophylaxis the number and rate of breakthrough infections will be reported. If breakthrough infection occurs the type of salvage therapy and the outcome will also be documented. For patients receiving anidulafungin as treatment of a current episode of a fungal infection the primary efficacy outcome is defined as the proportion of patients alive at week six after inclusion in the study or at the time that a patient is censored. A second evaluation of survival will be done at week 12. Reason of death will be analyzed according to toxicity of study drug and progression of IFI, respectively.

The efficacy outcome will be categorized into the following:

Success:

Complete response: Survival within the prespecified period of observation, resolution of all attributable symptoms and signs of disease and radiological abnormalities, and mycological evidence of eradication of disease.

Partial response: Survival within the prespecified period of observation, improvement in attributable symptoms and signs of disease and radiological abnormalities, and evidence of clearance of cultures or reduction of fungal burden, as assessed by a quantitative and validated laboratory marker.

Failure: Stable response: Survival within the prespecified period of observation and minor or no improvement in fungal disease, but no evidence of progression, as determined on the basis of a composite of clinical, radiological, and mycological criteria.

Progression: Evidence of progressive fungal disease based on a composite of clinical, radiological, and mycological criteria.

Death: Death during the prespecified period of evaluation, regardless of attribution.

Survival data (overall mortality and attributable mortality, if applicable) for all patients and the time-to-negativity of a blood culture will be reported in this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years) with a hematologic disorder AND an indication for IFI prophylaxis or therapy, but a relative contraindication for azoles or polyenes due to hepatic or renal dysfunction*, are scheduled to receive anidulafungin for one of the following specific indications:
* Need for primary antifungal prophylaxis in patients with Acute leucaemia/MDS during induction, reinduction or consolidation chemotherapy (who are expected to become neutropenic for at least 10 days) OR after allogenic HSCT with GvHD (at least grade II or more - systemic steroid treatment required)
* Need for secondary antifungal prophylaxis in patients with the history of a proven or probable invasive fungal infection who are expected to become neutropenic during induction, reinduction or consolidation chemotherapy
* Indication for treatment of proven**, probable or possible fungal infection:

  * Neutropenic patients with fever resistant to antibiotics (empirical use)
  * Neutropenic patients with fever resistant to antibiotics and additive laboratory or imaging signs of IFI (preemptive use)
  * Patients who failed other antifungal therapy due to intolerance or progressive infection

Exclusion Criteria:

* Absence of written informed consent
* Female patients who are pregnant or lactating
* Use of anidulafungin within 30 days prior to study
* Known hypersensitivity to anidulafungin
* Proven IFI with pathogen of known resistance to echinocandins (e.g. zygomycetes)
* Life expectancy less than 1 month
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Safety: incidence of (serious)adverse events and changes of important laboratory parameters (in particular liver and renal function parameters) with clinical impact will be reported. | day 1-5, 10 , end of treatment and study.

SECONDARY OUTCOMES:
pharmacokinetics and efficacy: As prophylaxis: the number of breakthrough infections. As treatment: complete and partial response rate (success); stable, progression and death (Failure) | day 5 (pharmacokinetics), end of treatment, week 6 and 12 (efficacy)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Girschikofsky, MD, Study Chair — Elisabethinen hospital Linz GmbH
Locations (1):
- Elisabethinen hospital, Linz, Upper Austria, Austria

REFERENCES:
- [Background] Damle BD, Dowell JA, Walsky RL, Weber GL, Stogniew M, Inskeep PB. In vitro and in vivo studies to characterize the clearance mechanism and potential cytochrome P450 interactions of anidulafungin. Antimicrob Agents Chemother. 2009 Mar;53(3):1149-56. doi: 10.1128/AAC.01279-08. Epub 2008 Nov 24. PMID 19029327
- [Background] Krause DS, Reinhardt J, Vazquez JA, Reboli A, Goldstein BP, Wible M, Henkel T; Anidulafungin Invasive Candidiasis Study Group. Phase 2, randomized, dose-ranging study evaluating the safety and efficacy of anidulafungin in invasive candidiasis and candidemia. Antimicrob Agents Chemother. 2004 Jun;48(6):2021-4. doi: 10.1128/AAC.48.6.2021-2024.2004. PMID 15155194
- [Background] Pappas PG, Kauffman CA, Andes D, Benjamin DK Jr, Calandra TF, Edwards JE Jr, Filler SG, Fisher JF, Kullberg BJ, Ostrosky-Zeichner L, Reboli AC, Rex JH, Walsh TJ, Sobel JD; Infectious Diseases Society of America. Clinical practice guidelines for the management of candidiasis: 2009 update by the Infectious Diseases Society of America. Clin Infect Dis. 2009 Mar 1;48(5):503-35. doi: 10.1086/596757. PMID 19191635
- [Background] Reboli AC, Rotstein C, Pappas PG, Chapman SW, Kett DH, Kumar D, Betts R, Wible M, Goldstein BP, Schranz J, Krause DS, Walsh TJ; Anidulafungin Study Group. Anidulafungin versus fluconazole for invasive candidiasis. N Engl J Med. 2007 Jun 14;356(24):2472-82. doi: 10.1056/NEJMoa066906. PMID 17568028
- [Background] De Pauw B, Walsh TJ, Donnelly JP, Stevens DA, Edwards JE, Calandra T, Pappas PG, Maertens J, Lortholary O, Kauffman CA, Denning DW, Patterson TF, Maschmeyer G, Bille J, Dismukes WE, Herbrecht R, Hope WW, Kibbler CC, Kullberg BJ, Marr KA, Munoz P, Odds FC, Perfect JR, Restrepo A, Ruhnke M, Segal BH, Sobel JD, Sorrell TC, Viscoli C, Wingard JR, Zaoutis T, Bennett JE; European Organization for Research and Treatment of Cancer/Invasive Fungal Infections Cooperative Group; National Institute of Allergy and Infectious Diseases Mycoses Study Group (EORTC/MSG) Consensus Group. Revised definitions of invasive fungal disease from the European Organization for Research and Treatment of Cancer/Invasive Fungal Infections Cooperative Group and the National Institute of Allergy and Infectious Diseases Mycoses Study Group (EORTC/MSG) Consensus Group. Clin Infect Dis. 2008 Jun 15;46(12):1813-21. doi: 10.1086/588660. PMID 18462102
- [Background] Segal BH, Herbrecht R, Stevens DA, Ostrosky-Zeichner L, Sobel J, Viscoli C, Walsh TJ, Maertens J, Patterson TF, Perfect JR, Dupont B, Wingard JR, Calandra T, Kauffman CA, Graybill JR, Baden LR, Pappas PG, Bennett JE, Kontoyiannis DP, Cordonnier C, Viviani MA, Bille J, Almyroudis NG, Wheat LJ, Graninger W, Bow EJ, Holland SM, Kullberg BJ, Dismukes WE, De Pauw BE. Defining responses to therapy and study outcomes in clinical trials of invasive fungal diseases: Mycoses Study Group and European Organization for Research and Treatment of Cancer consensus criteria. Clin Infect Dis. 2008 Sep 1;47(5):674-83. doi: 10.1086/590566. PMID 18637757
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009